CLINICAL TRIAL: NCT00313573
Title: TeleCare Management of Pain and Depression in Cancer
Brief Title: Telemedicine or Standard Care in Treating Patients With Depression and/or Pain Caused By Cancer
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Indiana University Melvin and Bren Simon Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Kurt Kroenke, Regenstrief Institute, Incorporated
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized
Other Study IDs: CDR0000466348; IUMC-051009
Record Dates: First submitted 2006-04-11; First posted 2006-04-12 (Estimated); Last update posted 2013-09-20 (Estimated); Status verified 2009-05

CONDITIONS: Depression; Pain; Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific; pain; depression
MeSH Terms: conditions — Depression; Pain | interventions — Analgesia; Psychiatric Rehabilitation

INTERVENTIONS:
Procedure: management of therapy complications
Procedure: pain therapy
Procedure: psychosocial assessment and care
Procedure: quality-of-life assessment

SUMMARY:
RATIONALE: Telemedicine may help in the treatment of depression and/or pain caused by cancer. It is not yet known whether telemedicine is more effective than standard care in treating depression and/or pain caused by cancer.

PURPOSE: This phase III randomized clinical trial is studying telemedicine to see how well it works compared to standard care in treating patients with depression and/or pain caused by cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Compare the effectiveness of a state-wide, telemedicine intervention with standard care in cancer patients with clinical depression and/or cancer-related pain.
* Compare improvement in clinical depression and/or cancer-related pain in patients undergoing these interventions.

Secondary

* Compare health-related quality of life, functional status, and patient satisfaction with treatment in patients undergoing these interventions.
* Compare the economic benefits of these interventions in these patients.

OUTLINE: This is a randomized, longitudinal, multicenter study. Patients are stratified according to study site and type of symptom (pain only vs depression only vs pain and depression). Patients are randomized to 1 of 2 treatment arms.

* Arm I (standard care): Patients receive treatment for pain, depression, and other symptoms from their oncologist.
* Arm II (telemedicine intervention): Patients undergo automated, home-based symptom monitoring either by telephone or the Internet, depending on preference, coupled with telephonic care management by a clinical specialist. Patients complete questionnaires via the Internet or undergo standardized interviews via telephone measuring depression, pain, quality of life, and other patient-reported variables twice weekly for approximately 1 month, once weekly for 2 months, twice a month for 3 months, and then once a month for 6 months. A clinical specialist trained in treating the symptoms of pain and depression also contacts the patient by phone to assess symptom severity and initiate treatment. A follow-up call is made at 1-2 weeks to assess symptom severity, adherence, and adverse effects. Patients with depression receive 2 additional follow-up calls in the first 12 weeks. The clinical specialist also calls the patient when automated monitoring indicates inadequate symptom improvement or side effects, or the patient requests to be contacted. The clinical specialist works with the patient's regular doctor in adjusting medicines and treatment for symptoms as needed. Patients who do not complete their scheduled assessments receive an automated call or e-mail message reminding them to complete the symptoms questionnaires. Patients who do not respond to this reminder within 24 hours are contacted by the clinical specialist.

In both arms, patients are interviewed at baseline, 1, 3, 6, and 12 months. Patients are asked questions about pain, depression, other physical and emotional symptoms, work activities, quality of life, and satisfaction with treatment.

PROJECTED ACCRUAL: A total of 480 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of cancer AND 1 or both of the following:

  * Clinical depression

    * Depression must be of at least moderate severity (PHQ-9 score ≥ 10)

      * Depressed mood and/or anhedonia endorsed
    * No depression directly precipitated by cancer therapy for which depression is a well known side effect (e.g., interferon, corticosteroids)
  * Cancer-related pain

    * Pain must be at least moderate in severity (Brief Pain Inventory score ≥ 6), persisted despite using ≥ 2 analgesics, and cancer-related
    * If the only pain is due to a pre-existing condition (e.g., migraine, headache, arthritis, etc), the patient may not be eligible

PATIENT CHARACTERISTICS:

* Life expectancy ≥ 6 months
* Must speak English
* Not pregnant
* Fertile patients must use effective contraception
* No moderately severe cognitive impairment
* No schizophrenia or other psychosis
* No disability claim currently being adjudicated for pain

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* Not in hospice care

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 480 (Estimated)
Dates: Start 2006-02; Primary Completion 2010-01 (Estimated)

PRIMARY OUTCOMES:
Compare efficacy of 3-component model telemedicine intervention to standard care in terms of depression and pain at baseline and 1, 3, 6, and 12 months

SECONDARY OUTCOMES:
Health-related quality of life at baseline and 1, 3, 6, and 12 months
Cost-effectiveness of care at baseline and 1, 3, 6, and 12 months
Treatment satisfaction at baseline and 1, 3, 6, and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Kurt Kroenke, MD, Study Chair — Regenstrief Institute, Incorporated
Locations (17):
- United States (17):
  - Community Cancer Center at Community Hospital of Anderson, Anderson, Indiana
  - Community Cancer Care at Bedford Oncology Specialty Clinic, Bedford, Indiana
  - Columbus Regional Hospital Cancer Center, Columbus, Indiana
  - Community Cancer Care at Putnam County Hospital, Greencastle, Indiana
  - Community Cancer Care at Decatur County Hospital, Greensburg, Indiana
  - Regenstrief Institute, Incorporated, Indianapolis, Indiana
  - Community Cancer Care, Indianapolis, Indiana
  - Veterans Affairs Medical Center - Indianapolis, Indianapolis, Indiana
  - William N. Wishard Memorial Hospital, Indianapolis, Indiana
  - Methodist Cancer Center at Methodist Hospital, Indianapolis, Indiana
  - Community Regional Cancer Care at Community Hospital East, Indianapolis, Indiana
  - Community Regional Cancer Care at Community Hospital North, Indianapolis, Indiana
  - Community Cancer Care at Howard Regional Health System, Kokomo, Indiana
  - Community Cancer Care at King's Daughters' Hospital, Madison, Indiana
  - Schneck Medical Center, Seymour, Indiana
  - Community Cancer Care at Perry County Hospital, Tell City, Indiana
  - Community Cancer Care at Tipton County Memorial Hospital, Tipton, Indiana

REFERENCES:
- [Result] Brown LF, Kroenke K, Theobald DE, Wu J, Tu W. The association of depression and anxiety with health-related quality of life in cancer patients with depression and/or pain. Psychooncology. 2010 Jul;19(7):734-41. doi: 10.1002/pon.1627. PMID 19777535
- [Result] Kroenke K, Theobald D, Wu J, Norton K, Morrison G, Carpenter J, Tu W. Effect of telecare management on pain and depression in patients with cancer: a randomized trial. JAMA. 2010 Jul 14;304(2):163-71. doi: 10.1001/jama.2010.944. PMID 20628129
- [Result] Kroenke K, Zhong X, Theobald D, Wu J, Tu W, Carpenter JS. Somatic symptoms in patients with cancer experiencing pain or depression: prevalence, disability, and health care use. Arch Intern Med. 2010 Oct 11;170(18):1686-94. doi: 10.1001/archinternmed.2010.337. PMID 20937930
- [Derived] He A, Kroenke K, Stump T, Monahan PO, Connors J, Chernyak Y, Musey P. The patient health questionnaire somatization-anxiety-depression scale: Validation of the PHQ-SAD in 4 clinical trials. J Affect Disord. 2026 Apr 1;398:120906. doi: 10.1016/j.jad.2025.120906. Epub 2025 Dec 21. PMID 41436014
- [Derived] Cohee AA, Kroenke K, Vachon E, Wu J, Tu W, Johns SA. Predictors of depression outcomes in adults with cancer: A 12 month longitudinal study. J Psychosom Res. 2020 Sep;136:110169. doi: 10.1016/j.jpsychores.2020.110169. Epub 2020 Jun 11. PMID 32559503
- [Derived] Kroenke K, Wu J, Yu Z, Bair MJ, Kean J, Stump T, Monahan PO. Patient Health Questionnaire Anxiety and Depression Scale: Initial Validation in Three Clinical Trials. Psychosom Med. 2016 Jul-Aug;78(6):716-27. doi: 10.1097/PSY.0000000000000322. PMID 27187854
- [Derived] Choi Yoo SJ, Nyman JA, Cheville AL, Kroenke K. Cost effectiveness of telecare management for pain and depression in patients with cancer: results from a randomized trial. Gen Hosp Psychiatry. 2014 Nov-Dec;36(6):599-606. doi: 10.1016/j.genhosppsych.2014.07.004. Epub 2014 Jul 19. PMID 25130518
- [Derived] Hayano J, Carney RM, Watanabe E, Kawai K, Kodama I, Stein PK, Watkins LL, Freedland KE, Blumenthal JA. Interactive associations of depression and sleep apnea with adverse clinical outcomes after acute myocardial infarction. Psychosom Med. 2012 Oct;74(8):832-9. doi: 10.1097/PSY.0b013e31826d2c81. Epub 2012 Sep 28. PMID 23023681
- [Derived] Wang HL, Kroenke K, Wu J, Tu W, Theobald D, Rawl SM. Predictors of cancer-related pain improvement over time. Psychosom Med. 2012 Jul-Aug;74(6):642-7. doi: 10.1097/PSY.0b013e3182590904. Epub 2012 Jun 28. PMID 22753637
- [Derived] Dube P, Kurt K, Bair MJ, Theobald D, Williams LS. The p4 screener: evaluation of a brief measure for assessing potential suicide risk in 2 randomized effectiveness trials of primary care and oncology patients. Prim Care Companion J Clin Psychiatry. 2010;12(6):PCC.10m00978. doi: 10.4088/PCC.10m00978blu. PMID 21494337